CLINICAL TRIAL: NCT01533012
Title: Initial Positioning of Left Sided Double Lumen Endobronchial Tubes Using Peak Inspiratory Pressures Difference Between Two Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2011-0619
Record Dates: First submitted 2012-02-07; First posted 2012-02-15 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pressure difference (Experimental): Peak inspiratory pressures difference between two lungs
  Interventions: Procedure: Pressure difference
- FOB evaluation (No Intervention): FOB evaluation for the optimal position of tubes

INTERVENTIONS:
Procedure: Pressure difference — Peak inspiratory pressures difference between two lungs
  Arms: Pressure difference

SUMMARY:
The purpose of this study is to investigate a performance of initial positioning of left sided double lumen endobronchial tubes using peak inspiratory pressures difference between two lungs.

DETAILED DESCRIPTION:
If both lungs have relatively equal volumes and the double lumen tube is in a satisfactory position, peak inspiratory pressure between two lungs is similar or equal when each lumen is sequentially clamped while ventilating each lung with the same tidal volume. We are going to investigate a performance of this method by fiberoptic bronchoscopy view and depth of double lumen tube, and compare with an conventional auscultation method.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I, II
* Use of double lumen tube
* Normal preoperative pulmonary function study

Exclusion Criteria:

* COPD
* Restrictive lung disease
* CAOD
* Unstable hemodynamic status
* Peak inspiratory pressure > 30 mm Hg (Two lung ventilation)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-10-25 (Actual); Study Completion 2012-10-25 (Actual)

PRIMARY OUTCOMES:
Fiberoptic bronchoscopy view | within 5 min after intubation
  1. aucsultation under manual ventilation -> fiberopric bronchoscopy view check
  2. peak inspiratory pressure difference under mechanical ventilation -> fiberoptic bronchoscopy view check

SECONDARY OUTCOMES:
depth of double lumen tube | within 5 min after checking fiberopitics
  1. aucsultation under manual ventilation -> A depth of DLT (incisor)
  2. peak inspiratory pressure difference under mechanical ventilation -> A depth of DLT (incisor)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine , Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Choi YS, Shin S, Cho JS, Nam DJ, Oh YJ. Positioning of double-lumen tubes based on the minimum peak inspiratory pressure difference between the right and left lungs in short patients: a prospective observational study. Eur J Anaesthesiol. 2014 Mar;31(3):137-42. doi: 10.1097/EJA.0b013e328364c3a7. PMID 24047768